CLINICAL TRIAL: NCT07330908
Title: Impact of Different Norepinephrine Doses on Accuracy of Peripheral Perfusion Index in Predicting Tissue Perfusion in Septic Shock Patients
Brief Title: Different Norepinephrine Doses on Accuracy of Peripheral Perfusion Index in Predicting Tissue Perfusion in Septic Shock Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Abdelghafar Elbaghdady, Resident, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264MS735/11/24
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock; Peripheral Perfusion Index
Keywords: Norepinephrine; Peripheral Perfusion Index; Septic Shock; Tissue Perfusion
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients will receive norepinephrine <0.15 µg/kg/minute
  Interventions: Drug: Group I: Patients will receive norepinephrine <0.15 µg/kg/min
- Group II (Experimental): Patients will receive norepinephrine ≥ 0.15 µg/kg/minutes
  Interventions: Drug: Group II: Patients will receive norepinephrine ≥ 0.15 µg/kg/min

INTERVENTIONS:
Drug: Group I: Patients will receive norepinephrine <0.15 µg/kg/min — Patients will receive norepinephrine <0.15 µg/kg/min
  Arms: Group I
Drug: Group II: Patients will receive norepinephrine ≥ 0.15 µg/kg/min — Patients will receive norepinephrine ≥ 0.15 µg/kg/min
  Arms: Group II

SUMMARY:
This study aims to evaluate the impact of different norepinephrine doses on the accuracy of the peripheral perfusion index in predicting tissue perfusion in septic shock patients.

Primary outcome:

* Correlation between peripheral perfusion index

Secondary outcomes:

* Peripheral perfusion index accuracy to predict the tissue perfusion .
* Peripheral perfusion index accuracy to predict mortality.

DETAILED DESCRIPTION:
Septic shock is a common cause of intensive care unit admission and one of the major causes of death among intensive care unit inpatients.

It is a complex critical condition associated with a reported mortality rate of up to 30% to 40%.

. It is the most severe form of sepsis with concomitant hemodynamic failure and immune, inflammatory, and metabolic disorders. The resulting circulatory shock finally leads to an alteration of tissue perfusion, causing organ failures and associated poor outcomes.

An essential step in managing patients with septic shock is to increase systemic and regional/microcirculatory flow. Increasing arterial blood pressure with vasopressors when patients are hypotensive improves the input pressure that drives organ perfusion. Therefore, maintaining organ perfusion in the time course of septic shock is a fundamental goal.

Norepinephrine is a commonly used vasopressor in the management of septic shock. It increases vascular tone and blood pressure, thereby improving systemic perfusion. However, excessive norepinephrine dosing is associated with the risk of extreme vasoconstriction, tissue hypoperfusion, and increased mortality. Peripheral and regional tissue perfusion in patients with septic shock have been extensively studied over the last decade. Indeed, several authors have emphasized the potential benefits of monitoring microcirculatory and regional perfusion parameters to better guide the resuscitation of these patients and give a prognosis. The peripheral perfusion index ,which is defined as the ratio of the pulsatile to non-pulsatile component of the pulse oximetry plethysmograph (peripheral perfusion index = pulsatile signal/ non-pulsatile signal), is used as a simple and accurate indicator of the pulsation intensity of peripheral arterioles .

We hypothesize that peripheral perfusion index could accurately predict tissue perfusion at different doses of norepinephrine in septic shock patients. This study aims to evaluate the impact of different norepinephrine doses on the accuracy of the peripheral perfusion index in predicting tissue perfusion in septic shock patients.

Primary outcome:

* Correlation between peripheral perfusion index

Secondary outcomes:

* Peripheral perfusion index accuracy to predict the tissue perfusion .
* Peripheral perfusion index accuracy to predict mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Both sexes.
* Septic shock patients requiring norepinephrine infusion at dose <0.25 µg/kg/min to achieve mean arterial pressure (Mean arterial blood pressure ≥ 65 mm Hg).

Exclusion Criteria:

* Patients fail to achieve Mean arterial blood ≥ 65 mm Hg or need norepinephrine dose ≥0.25 µg /kg/min.
* Pregnancy.
* Diabetes mellitus.
* Tissue edema.
* Respiratory diseases affecting gas exchange, such as asthma and Chronic Obstructive Pulmonary Disease.
* Sever hypoxemia or hypercarbia.
* Core temperature < 36 ᴼc.
* Body mass index ≥35 kg/m2
* Cardiovascular diseases and pulmonary edema

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Peripheral Perfusion Index and ( Central venous oxygen saturation , and lactate clearance). | Before initiation of vasopressor therapy, 5 minutes, 30 minutes, 1 hour, 2 hours, and 6 hours post-initiation of vasopressor therapy

SECONDARY OUTCOMES:
Mean arterial blood pressure | Before the initiation of vasopressor therapy, 5 minutes, 30 minutes,, 1 hour, 2 hours, and 6 hours after the initiation of vasopressor therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It will be provided when required
Supporting Information: Study Protocol, ICF